CLINICAL TRIAL: NCT01990534
Title: A Single-arm Study of Brentuximab Vedotin in Patients With Relapsed or Refractory Hodgkin Lymphoma Who Are Not Suitable for Stem Cell Transplantation or Multiagent Chemotherapy
Brief Title: A Study of Brentuximab Vedotin in Participants With Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25007; 2013-000232-10 (EudraCT Number); U1111-1154-2250 (Registry Identifier: WHO); NMRR-13-1246-18099 (Registry Identifier: NMRR); REec-2014-0619 (Registry Identifier: REec)
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Hodgkin Lymphoma
Keywords: Lymphoma; Hodgkin; Relapsed; Refractory; Antigens, CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; Monomethyl auristatin E; Drug Therapy; Immunotherapy; Hematologic Diseases; Additional Relevant MeSH terms:; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Hodgkin; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, B-Cell; Lymphoma, T-Cell; Immunologic Factors; Physiological Effects of Drugs; Pharmacologic Actions
MeSH Terms: conditions — Hodgkin Disease; Lymphoma; Recurrence; Hematologic Diseases; Lymphoma, Large B-Cell, Diffuse; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, B-Cell; Lymphoma, T-Cell | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin 1.8 mg/kg (Experimental): Brentuximab vedotin 1.8 mg/kg, 30-minute intravenous (IV) infusion, Day 1 in every 3-week cycle, until there is evidence of disease progression or unacceptable toxicity occurs (Up to 16 cycles). The dose could be decreased or delayed or discontinued in participants who develop treatment-associated non-hematologic, hematologic toxicity or peripheral neuropathy to brentuximab vedotin.
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab vedotin IV infusion
  Other Names: SGN-35; ADCETRIS

SUMMARY:
This phase 4, single-arm, open-label, multicenter study is designed to evaluate the efficacy and safety of brentuximab vedotin as a single agent in adult participants with histologically confirmed CD30+ relapsed or refractory classical Hodgkin Lymphoma who have not received a prior stem cell transplantation (SCT) and are considered to be not suitable for SCT or multiagent chemotherapy at the time of study entry.

DETAILED DESCRIPTION:
The drug being tested in this study is called brentuximab vedotin. Brentuximab vedotin is being tested to treat people who have relapsed or refractory Hodgkin Lymphoma. This study will look at the overall response of people who took brentuximab vedotin.

The study will enroll 60 patients. Participants received:

• Brentuximab vedotin 1.8 mg/kg

This multicenter trial is being conducted worldwide. The overall time to participate in this study is approximately 6 to 7 years. Participants will make multiple visits to the clinic, and will be contacted by telephone every 3 months for 18 months after the end of treatment (EOT) for follow-up assessment of overall survival and then every 6 months until death, study closure, or 5 years after enrollment of the last participant.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to be enrolled in the study:

1. Male or female participants 18 years or older, with relapsed or refractory classical Hodgkin lymphoma (HL), who have previously received at least 1 prior systemic chemotherapeutic regimen
2. Not suitable for stem cell transplantation (SCT) or multiagent chemotherapy, according to 1 of the following criteria:

   * Disease progression within 90 days of the earliest date of complete remission (CR) or complete remission unconfirmed (CRu) after the end of treatment with multiagent chemotherapeutic regimens and/or radiotherapy
   * Progressive disease during frontline multiagent chemotherapy
   * Disease relapse after treatment with at least 2 chemotherapeutic regimens, including any salvage treatments
3. Bidimensional measurable disease
4. An Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
5. Female participants who are postmenopausal for at least 1 year before the screening visit, surgically sterile, or agree to practice 2 effective methods of contraception at the same time, or agree to practice true abstinence.
6. Male participants who agree to practice effective barrier contraception during the entire study treatment period through 6 months after the last dose of study drug or agree to practice true abstinence.
7. Clinical laboratory values as specified in the study protocol.

Exclusion Criteria:

Participants who meet any of the following exclusion criteria are not to be enrolled in the study:

1. Previous treatment with brentuximab vedotin
2. Previously received an autologous stem cell transplantation (ASCT) or alloSCT
3. Known cerebral/meningeal disease, including signs or symptoms suggestive of progressive multifocal leukoencephalopathy (PML), or any history of PML.
4. Female participants who are lactating and breastfeeding or pregnant.
5. Known human immunodeficiency virus (HIV).
6. Known hepatitis B surface antigen positive, or known or suspected active hepatitis C infection.
7. Grade 2 or higher peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2016-03-24 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (18):
- Czechia (2):
  - Prague, Prague
  - Brno
- Germany (2):
  - Heidelberg, Baden-Wurttemberg
  - Cologne
- Malaysia (3):
  - George Town, Pulau Pinang
  - Ampang, Selangor
  - Kuala Lumpur
- Poland (3):
  - Gdansk
  - Krakow
  - Warsaw
- Spain (2):
  - Pamplona, Navarre
  - Madrid
- Thailand (3):
  - Bangkoknoi, Bangkok
  - Patumwan, Bangkok
  - Ratchathewi, Bangkok
- Turkey (Türkiye) (3):
  - Izmir, Bornova
  - Ankara
  - Izmir

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 investigative sites in Czech Republic, Germany, Malaysia, Poland, Spain, Thailand and Turkey, from 14 March 2014 to 12 March 2020.
Pre-assignment Details: Participants with a diagnosis of relapsed or refractory Hodgkin Lymphoma were enrolled in 1 treatment group to receive brentuximab vedotin 1.8 mg/kg, 30-minute intravenous (IV) infusion on Day 1 of every 3-week cycle and were followed for progression free survival (PFS) and overall survival (OS) up to the End of study (approximately 6 years).
Groups:
- Brentuximab Vedotin 1.8 mg/kg: Brentuximab vedotin 1.8 mg/kg, 30-minute IV infusion, Day 1 of every 3-week cycle, until there is evidence of disease progression or unacceptable toxicity occurs (Up to 16 cycles). The dose could be decreased or delayed or discontinued in participants who develop treatment-associated non-hematologic toxicity, hematologic toxicity or peripheral neuropathy to brentuximab vedotin.
Period: Overall Study
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Started | 60
Completed | 25
Not Completed | 35
Not completed — Death | 22
Not completed — Progressive disease | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal of Informed Consent | 2
Not completed — Symptomatic Deterioration | 1
Not completed — Withdrawal by Subject | 3
Not completed — Reason not Specified | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all enrolled participants who received at least 1 dose of brentuximab vedotin.
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Czech Republic | 3
  Germany | 2
  Malaysia | 8
  Poland | 26
  Spain | 2
  Thailand | 10
  Turkey | 9
Baseline Height [Mean (Standard Deviation); unit: cm] | 171.0 (9.66)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 70.3 (19.41)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = weight (kg)/[height (m)^2]
  kg/m^2 | 23.864 (5.4085)

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the percentage of participants with complete remission (CR) or partial remission (PR) as assessed by an independent review facility (IRF) using International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma. CR is defined as the disappearance of all evidence of disease and PR is defined as regression of measurable disease and no new sites.
Time Frame: Baseline until disease progression, death or end of study (EOS) (Up to 24 months)
Population: Intent-to-Treat (ITT) Population included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
percentage of participants | 50 [37 to 63]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time in months from the date of first documentation of a CR or PR response to the date of first documentation of tumor progression or progressive disease (PD) per IRF assessment according to IWG criteria. CR is defined as the disappearance of all evidence of disease. PR is defined as regression of measurable disease and no new sites. PD is defined as any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: From first documented complete or partial remission until disease progression (Up to 24 months)
Population: ITT Population included all participants who were enrolled in the study. DOR was censored on the date of last disease assessment documenting absence of PD for those that were lost to follow-up, withdrew consent, started a new anticancer therapy other than stem cell transplantation (SCT), or discontinued treatment due to undocumented PD after last disease assessment. All responders were evaluated in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 30
months | 4.6 [3.42 to 7.85]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as time in months from start of study treatment to first documentation of objective tumor progression per IRF assessment or up to death due to any cause, whichever occurs first.
Time Frame: Baseline until disease progression, death or end of treatment (EOT), and then every 3 months up to approximately 6 years
Population: ITT Population included all participants who were enrolled in the study. For a participant that has not progressed and has not died, PFS is censored at the last response assessment that is SD or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
months | 4.8 [2.96 to 5.32]

4. Secondary Outcome: Complete Remission Rate
Description: Complete remission rate is defined as percentage of participants with CR per IRF response assessment based on IWG criteria are reported. CR is defined as the disappearance of all evidence of disease.
Time Frame: Baseline until disease progression, death or EOS (Up to approximately 6 years)
Population: ITT Population included all participants who were enrolled in the study. In the absence of confirmation of death, survival time is censored at the last date the participant is known to be alive, including study closure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
percentage of participants | 13 [6 to 25]

5. Secondary Outcome: Duration of Complete Remission
Description: Duration of CR is defined as the time from the date of first documentation of a CR or to the date of first documentation of tumor progression or progressive disease (PD) per IRF assessment according to IWG criteria. CR is defined as the disappearance of all evidence of disease and PD is defined as any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: From first documented complete remission until disease progression (up to approximately 6 years)
Population: ITT Population included all participants who were enrolled in the study. Duration of complete remission was censored on the date of last disease assessment documenting absence of PD for those that were lost to follow-up, withdrew consent, started a new anticancer therapy other than SCT, or discontinued treatment due to undocumented PD after last disease assessment. Only participants with CR were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 8
months | 6.1 [2.10 to NA] — Upper limit of CI was not estimable due to the low number of participants with events.

6. Secondary Outcome: Overall Survival (OS)
Description: OS is the time in months from start of study treatment to date of death due to any cause.
Time Frame: Every 3 months for 18 months after EOT, thereafter, every 6 months until the sooner of death, study closure, or 5 years after enrollment of the last participant (up to approximately 6 years)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
months | NA [NA to NA] — Median and 95% confidence interval (CI) was not estimable due to the low number of participants with events.

7. Secondary Outcome: Percentage of Participants Who Received Hematopoietic SCT
Time Frame: Baseline up to EOS (up to approximately 6 years)
Population: ITT Population included all participants who were enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
percentage of participants | 53

8. Secondary Outcome: Number of Participants With Adverse Events (AEs), Drug-Related AEs, Grade 3 or Higher AEs, Serious Adverse Events (SAEs), Drug-Related SAEs and Grade 3 or Higher SAEs
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A SAE a serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. AE severity was graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. AEs Grade 3 and higher are severe.
Time Frame: From first dose through 30 days after the last dose of study medication (Up to 24 months)
Population: Safety Population was defined as all enrolled participants who received at least one dose of brentuximab vedotin.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
Participants
  Any AEs | 52
  Grade 3 or higher AEs | 21
  Drug-related AEs | 41
  Drug-related Grade 3 or higher AEs | 11
  SAEs | 11
  Drug-related SAEs | 3

9. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Values Reported as AEs
Description: Abnormal clinical laboratory values (serum chemistry and hematology) were reported as AEs if they were considered by the investigator to be a clinically significant change from Baseline or led to premature discontinuation of study treatment, dose modification, or other therapeutic intervention.
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 24 months)
Population: Safety Population was defined as all enrolled participants who received at least one dose of brentuximab vedotin.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
Participants
  Neutrophil count decreased | 2
  Lymphocyte count decreased | 1
  Alanine aminotransferase increased | 2
  Aspartate aminotransferase increased | 2
  Gamma-glutamyltransferase increased | 1
  Blood thyroid stimulating hormone increased | 1
  Platelet count decreased | 1
  Haemoglobin decreased | 1
  Blood alkaline phosphatase increased | 1
  Blood lactate dehydrogenase increased | 1

10. Secondary Outcome: Antibody-drug Conjugate (ADC) Serum Concentrations
Description: Blood samples were collected and tested for serum concentrations of brentuximab vedotin antibody-drug conjugate.
Time Frame: Cycle 1 pre-dose and 10 minutes, 24 hours and 336 hours post-dose; Cycle 2 pre-dose and 10 minutes post-dose; Cycle 3 pre-dose and 10 minutes, 24 hours and 336 hours post-dose; Cycle 4 to 16 pre-dose and 10 minutes post-dose; EOT (Up to 24 months)
Population: Pharmacokinetic (PK)-evaluable Population was defined as participants with sufficient dosing and PK data to reliably estimate PK parameters. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
ng/mL
  Cycle 1 Day 1, Pre-Dose: number analyzed (Participants) | 59
  Cycle 1 Day 1, Pre-Dose | 0.00 (0.000)
  Cycle 1 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 58
  Cycle 1 Day 1, 10 minutes Post-Dose | 35504.65 (10226.104)
  Cycle 1 Day 2, 24 hours Post-Dose: number analyzed (Participants) | 59
  Cycle 1 Day 2, 24 hours Post-Dose | 14517.67 (4481.312)
  Cycle 1 Day 15, 336 hours Post-Dose: number analyzed (Participants) | 55
  Cycle 1 Day 15, 336 hours Post-Dose | 1410.43 (1946.525)
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 52
  Cycle 2 Day 1, Pre-Dose | 526.42 (350.467)
  Cycle 2 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 53
  Cycle 2 Day 1, 10 minutes Post-Dose | 37118.32 (11678.088)
  Cycle 3 Day 1, Pre-Dose: number analyzed (Participants) | 49
  Cycle 3 Day 1, Pre-Dose | 2283.30 (7552.322)
  Cycle 3 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 51
  Cycle 3 Day 1, 10 minutes Post-Dose | 35878.77 (12724.898)
  Cycle 3 Day 2, 24 hours Post-Dose: number analyzed (Participants) | 54
  Cycle 3 Day 2, 24 hours Post-Dose | 14737.82 (4512.358)
  Cycle 3 Day 15, 336 hours Post-Dose: number analyzed (Participants) | 46
  Cycle 3 Day 15, 336 hours Post-Dose | 1586.45 (680.955)
  Cycle 4 Day 1, Pre-Dose: number analyzed (Participants) | 51
  Cycle 4 Day 1, Pre-Dose | 1313.56 (2566.360)
  Cycle 4 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 51
  Cycle 4 Day 1, 10 minutes Post-Dose | 42915.34 (28221.764)
  Cycle 5 Day 1, Pre-Dose: number analyzed (Participants) | 43
  Cycle 5 Day 1, Pre-Dose | 1117.01 (637.637)
  Cycle 5 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 41
  Cycle 5 Day 1, 10 minutes Post-Dose | 36418.77 (10041.935)
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 37
  Cycle 6 Day 1, Pre-Dose | 1231.45 (714.383)
  Cycle 6 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 38
  Cycle 6 Day 1, 10 minutes Post-Dose | 39000.95 (12484.458)
  Cycle 7 Day 1, Pre-Dose: number analyzed (Participants) | 38
  Cycle 7 Day 1, Pre-Dose | 1285.91 (712.625)
  Cycle 7 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 36
  Cycle 7 Day 1, 10 minutes Post-Dose | 38814.82 (12471.299)
  Cycle 8 Day 1, Pre-Dose: number analyzed (Participants) | 22
  Cycle 8 Day 1, Pre-Dose | 1413.98 (782.391)
  Cycle 8 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 24
  Cycle 8 Day 1, 10 minutes Post-Dose | 39027.22 (9919.251)
  Cycle 9 Day 1, Pre-Dose: number analyzed (Participants) | 15
  Cycle 9 Day 1, Pre-Dose | 1277.18 (594.603)
  Cycle 9 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 14
  Cycle 9 Day 1, 10 minutes Post-Dose | 38359.15 (13421.064)
  Cycle 10 Day 1, Pre-Dose: number analyzed (Participants) | 11
  Cycle 10 Day 1, Pre-Dose | 1498.44 (754.721)
  Cycle 10 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 11
  Cycle 10 Day 1, 10 minutes Post-Dose | 39890.12 (5376.038)
  Cycle 11 Day 1, Pre-Dose: number analyzed (Participants) | 9
  Cycle 11 Day 1, Pre-Dose | 1511.35 (461.907)
  Cycle 11 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 9
  Cycle 11 Day 1, 10 minutes Post-Dose | 39132.17 (6316.541)
  Cycle 12 Day 1, Pre-Dose: number analyzed (Participants) | 10
  Cycle 12 Day 1, Pre-Dose | 1479.38 (397.816)
  Cycle 12 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 10
  Cycle 12 Day 1, 10 minutes Post-Dose | 39955.13 (7821.656)
  Cycle 13 Day 1, Pre-Dose: number analyzed (Participants) | 9
  Cycle 13 Day 1, Pre-Dose | 1423.56 (415.744)
  Cycle 13 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 9
  Cycle 13 Day 1, 10 minutes Post-Dose | 37609.69 (4563.601)
  Cycle 14 Day 1, Pre-Dose: number analyzed (Participants) | 8
  Cycle 14 Day 1, Pre-Dose | 1185.62 (422.664)
  Cycle 14 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 8
  Cycle 14 Day 1, 10 minutes Post-Dose | 38282.29 (10324.023)
  Cycle 15 Day 1, Pre-Dose: number analyzed (Participants) | 8
  Cycle 15 Day 1, Pre-Dose | 2279.42 (2919.545)
  Cycle 15 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 8
  Cycle 15 Day 1, 10 minutes Post-Dose | 39068.14 (7981.110)
  Cycle 16 Day 1, Pre-Dose: number analyzed (Participants) | 8
  Cycle 16 Day 1, Pre-Dose | 1452.23 (429.731)
  Cycle 16 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 8
  Cycle 16 Day 1, 10 minutes Post-Dose | 38414.73 (9427.315)
  End of Treatment: number analyzed (Participants) | 49
  End of Treatment | 1515.30 (6413.367)

11. Secondary Outcome: Serum Concentration of Total Antibodies (Conjugated and Unconjugated)
Description: Blood samples were collected and tested for conjugated and unconjugated antibodies.
Time Frame: as for outcome 10
Population: PK-evaluable Population was defined as participants with sufficient dosing and PK data to reliably estimate PK parameters. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
ng/mL
  Cycle 1 Day 1, Pre-Dose: number analyzed (Participants) | 58
  Cycle 1 Day 1, Pre-Dose | 0.00 (0.000)
  Cycle 1 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 57
  Cycle 1 Day 1, 10 minutes Post-Dose | 37329.59 (17724.247)
  Cycle 1 Day 2, 24 hours Post-Dose: number analyzed (Participants) | 57
  Cycle 1 Day 2, 24 hours Post-Dose | 23248.90 (8228.938)
  Cycle 1 Day 15, 336 hours Post-Dose: number analyzed (Participants) | 59
  Cycle 1 Day 15, 336 hours Post-Dose | 2791.49 (1413.452)
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 56
  Cycle 2 Day 1, Pre-Dose | 1254.86 (774.586)
  Cycle 2 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 54
  Cycle 2 Day 1, 10 minutes Post-Dose | 39801.87 (12914.837)
  Cycle 3 Day 1, Pre-Dose: number analyzed (Participants) | 54
  Cycle 3 Day 1, Pre-Dose | 2645.22 (5685.914)
  Cycle 3 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 52
  Cycle 3 Day 1, 10 minutes Post-Dose | 36461.28 (11144.634)
  Cycle 3 Day 2, 24 hours Post-Dose: number analyzed (Participants) | 50
  Cycle 3 Day 2, 24 hours Post-Dose | 27071.46 (8069.489)
  Cycle 3 Day 15, 336 hours Post-Dose: number analyzed (Participants) | 49
  Cycle 3 Day 15, 336 hours Post-Dose | 4033.28 (1760.094)
  Cycle 4 Day 1, Pre-Dose: number analyzed (Participants) | 52
  Cycle 4 Day 1, Pre-Dose\ | 2600.73 (2275.881)
  Cycle 4 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 50
  Cycle 4 Day 1, 10 minutes Post-Dose | 41823.31 (11761.223)
  Cycle 5 Day 1, Pre-Dose: number analyzed (Participants) | 43
  Cycle 5 Day 1, Pre-Dose | 2690.61 (1254.886)
  Cycle 5 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 42
  Cycle 5 Day 1, 10 minutes Post-Dose | 43786.57 (15470.979)
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 39
  Cycle 6 Day 1, Pre-Dose | 2806.17 (1021.877)
  Cycle 6 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 39
  Cycle 6 Day 1, 10 minutes Post-Dose | 44936.89 (13827.929)
  Cycle 7 Day 1, Pre-Dose: number analyzed (Participants) | 38
  Cycle 7 Day 1, Pre-Dose | 3889.94 (6201.351)
  Cycle 7 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 36
  Cycle 7 Day 1, 10 minutes Post-Dose | 41840.20 (12552.597)
  Cycle 8 Day 1, Pre-Dose: number analyzed (Participants) | 24
  Cycle 8 Day 1, Pre-Dose | 2932.19 (1089.138)
  Cycle 8 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 24
  Cycle 8 Day 1, 10 minutes Post-Dose | 42013.77 (12754.334)
  Cycle 9 Day 1, Pre-Dose: number analyzed (Participants) | 15
  Cycle 9 Day 1, Pre-Dose | 2959.26 (970.811)
  Cycle 9 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 14
  Cycle 9 Day 1, 10 minutes Post-Dose | 37300.95 (13442.910)
  Cycle 10 Day 1, Pre-Dose: number analyzed (Participants) | 11
  Cycle 10 Day 1, Pre-Dose | 3189.16 (1484.258)
  Cycle 10 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 11
  Cycle 10 Day 1, 10 minutes Post-Dose | 38910.05 (6169.552)
  Cycle 11 Day 1, Pre-Dose: number analyzed (Participants) | 10
  Cycle 11 Day 1, Pre-Dose | 3393.07 (1160.604)
  Cycle 11 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 10
  Cycle 11 Day 1, 10 minutes Post-Dose | 41238.25 (8081.750)
  Cycle 12 Day 1, Pre-Dose: number analyzed (Participants) | 10
  Cycle 12 Day 1, Pre-Dose | 3270.44 (965.895)
  Cycle 12 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 10
  Cycle 12 Day 1, 10 minutes Post-Dose | 37550.64 (12459.906)
  Cycle 13 Day 1, Pre-Dose: number analyzed (Participants) | 9
  Cycle 13 Day 1, Pre-Dose | 3406.00 (1067.414)
  Cycle 13 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 9
  Cycle 13 Day 1, 10 minutes Post-Dose | 35694.80 (3720.378)
  Cycle 14 Day 1, Pre-Dose: number analyzed (Participants) | 8
  Cycle 14 Day 1, Pre-Dose | 2723.01 (1286.457)
  Cycle 14 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 8
  Cycle 14 Day 1, 10 minutes Post-Dose | 40848.64 (8704.538)
  Cycle 15 Day 1, Pre-Dose: number analyzed (Participants) | 8
  Cycle 15 Day 1, Pre-Dose | 3111.63 (941.200)
  Cycle 15 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 8
  Cycle 15 Day 1, 10 minutes Post-Dose | 37091.56 (6644.258)
  Cycle 16 Day 1, Pre-Dose: number analyzed (Participants) | 8
  Cycle 16 Day 1, Pre-Dose | 3159.38 (1017.679)
  Cycle 16 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 8
  Cycle 16 Day 1, 10 minutes Post-Dose | 39266.07 (9358.163)
  End of Treatment: number analyzed (Participants) | 50
  End of Treatment | 2340.49 (6715.837)

12. Secondary Outcome: Monomethyl Auristatin E (MMAE) Serum Concentrations
Description: Blood samples were collected and tested for MMAE serum concentrations.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 60
pg/mL
  Cycle 1 Day 1, Pre-Dose: number analyzed (Participants) | 59
  Cycle 1 Day 1, Pre-Dose | 0.78 (5.976)
  Cycle 1 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 58
  Cycle 1 Day 1, 10 minutes Post-Dose | 591.09 (662.608)
  Cycle 1 Day 2, 24 hours Post-Dose: number analyzed (Participants) | 59
  Cycle 1 Day 2, 24 hours Post-Dose | 6056.44 (3850.457)
  Cycle 1 Day 15, 336 hours Post-Dose: number analyzed (Participants) | 59
  Cycle 1 Day 15, 336 hours Post-Dose | 746.12 (1123.502)
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 57
  Cycle 2 Day 1, Pre-Dose | 140.11 (111.036)
  Cycle 2 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 55
  Cycle 2 Day 1, 10 minutes Post-Dose | 539.38 (593.150)
  Cycle 3 Day 1, Pre-Dose: number analyzed (Participants) | 54
  Cycle 3 Day 1, Pre-Dose | 130.62 (84.152)
  Cycle 3 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 52
  Cycle 3 Day 1, 10 minutes Post-Dose | 484.88 (701.402)
  Cycle 3 Day 2, 24 hours Post-Dose: number analyzed (Participants) | 51
  Cycle 3 Day 2, 24 hours Post-Dose | 3076.75 (2330.510)
  Cycle 3 Day 15, 336 hours Post-Dose: number analyzed (Participants) | 49
  Cycle 3 Day 15, 336 hours Post-Dose | 442.63 (259.360)
  Cycle 4 Day 1, Pre-Dose: number analyzed (Participants) | 52
  Cycle 4 Day 1, Pre-Dose | 150.95 (123.841)
  Cycle 4 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 52
  Cycle 4 Day 1, 10 minutes Post-Dose | 497.20 (520.110)
  Cycle 5 Day 1, Pre-Dose: number analyzed (Participants) | 43
  Cycle 5 Day 1, Pre-Dose | 153.95 (123.337)
  Cycle 5 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 42
  Cycle 5 Day 1, 10 minutes Post-Dose | 392.50 (320.346)
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 39
  Cycle 6 Day 1, Pre-Dose | 158.89 (109.024)
  Cycle 6 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 39
  Cycle 6 Day 1, 10 minutes Post-Dose | 369.53 (260.871)
  Cycle 7 Day 1, Pre-Dose: number analyzed (Participants) | 38
  Cycle 7 Day 1, Pre-Dose | 185.91 (147.311)
  Cycle 7 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 37
  Cycle 7 Day 1, 10 minutes Post-Dose | 363.83 (237.883)
  Cycle 8 Day 1, Pre-Dose: number analyzed (Participants) | 24
  Cycle 8 Day 1, Pre-Dose | 136.37 (86.947)
  Cycle 8 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 24
  Cycle 8 Day 1, 10 minutes Post-Dose | 303.43 (202.351)
  Cycle 9 Day 1, Pre-Dose: number analyzed (Participants) | 15
  Cycle 9 Day 1, Pre-Dose | 142.30 (114.794)
  Cycle 9 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 14
  Cycle 9 Day 1, 10 minutes Post-Dose | 224.52 (159.833)
  Cycle 10 Day 1, Pre-Dose: number analyzed (Participants) | 11
  Cycle 10 Day 1, Pre-Dose | 100.78 (57.270)
  Cycle 10 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 11
  Cycle 10 Day 1, 10 minutes Post-Dose | 253.73 (113.311)
  Cycle 11 Day 1, Pre-Dose: number analyzed (Participants) | 10
  Cycle 11 Day 1, Pre-Dose | 158.09 (169.963)
  Cycle 11 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 10
  Cycle 11 Day 1, 10 minutes Post-Dose | 302.60 (175.869)
  Cycle 12 Day 1, Pre-Dose: number analyzed (Participants) | 10
  Cycle 12 Day 1, Pre-Dose | 175.02 (141.192)
  Cycle 12 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 10
  Cycle 12 Day 1, 10 minutes Post-Dose | 382.52 (428.255)
  Cycle 13 Day 1, Pre-Dose: number analyzed (Participants) | 9
  Cycle 13 Day 1, Pre-Dose | 146.76 (61.758)
  Cycle 13 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 9
  Cycle 13 Day 1, 10 minutes Post-Dose | 258.78 (108.871)
  Cycle 14 Day 1, Pre-Dose: number analyzed (Participants) | 8
  Cycle 14 Day 1, Pre-Dose | 82.13 (22.661)
  Cycle 14 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 8
  Cycle 14 Day 1, 10 minutes Post-Dose | 204.29 (121.162)
  Cycle 15 Day 1, Pre-Dose: number analyzed (Participants) | 8
  Cycle 15 Day 1, Pre-Dose | 133.78 (59.213)
  Cycle 15 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 8
  Cycle 15 Day 1, 10 minutes Post-Dose | 246.63 (98.399)
  Cycle 16 Day 1, Pre-Dose: number analyzed (Participants) | 8
  Cycle 16 Day 1, Pre-Dose | 163.39 (114.821)
  Cycle 16 Day 1, 10 minutes Post-Dose: number analyzed (Participants) | 8
  Cycle 16 Day 1, 10 minutes Post-Dose | 264.63 (103.269)
  End of Treatment: number analyzed (Participants) | 50
  End of Treatment | 139.72 (220.211)

13. Secondary Outcome: Number of Participants With Antitherapeutic Antibodies (ATA)
Description: Blood samples were collected to assess the immunogenicity of brentuximab vedotin (ATA development) using a laboratory test. Confirmed ATA-positive response was categorized as transient (defined as 1 or 2 post-Baseline confirmed ATA-positive responses) and persistent (defined as more than 2 post-Baseline confirmed ATA positive responses) and neutralizing ATA (nATA) status. The confirmed ATA-positive samples were assessed for ATA titer and delineated into having high or low titers.
Time Frame: Day 1 of every 3-week cycle up to 16 cycles and EOT (Up to 24 months)
Population: Participants from the Safety Population, all enrolled participants who received at least one dose of brentuximab vedotin, with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 56
Participants
  ATA Positive | 21
  Transient Positive | 17
  Persistently Positive | 4
  ATA Titer Low (≤25) | 21
  ATA Titer High (>25) | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 30 days post last dose of study drug (Up to 24 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
All-Cause Mortality (participants affected / at risk) | 22/60
Serious Adverse Events (participants affected / at risk) | 11/60
Other Adverse Events (participants affected / at risk) | 51/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.8 mg/kg (N=60)
Bronchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Serum sickness-like reaction (Immune system disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.8 mg/kg (N=60)
Anaemia (Blood and lymphatic system disorders) | 5
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Tachycardia (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Autoimmune thyroiditis (Endocrine disorders) | 1
Diplopia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 3
Catheter site inflammation (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Extravasation (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 11
Soft tissue inflammation (General disorders) | 1
Temperature regulation disorder (General disorders) | 1
Vaccination site pain (General disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Breast cellulitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 1
Coxsackie viral infection (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Pseudomonas infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 5
Viral infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Autonomic neuropathy (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 7
Polyneuropathy (Nervous system disorders) | 5
Somnolence (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Renal tubular disorder (Renal and urinary disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2013-07-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT01990534/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT01990534/SAP_001.pdf